CLINICAL TRIAL: NCT00998647
Title: Assessment of the Influence of Modified Ultrafiltration on Primary and Secondary Hemostasis in Cardiac Surgery Patients
Brief Title: Modified Ultrafiltration in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Christian Weber / Dr. med., Clinic for Anaesthesiology, Johann Wolfgang Goethe University Frankfurt
Other Study IDs: 370/08 MUF
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2009-10

CONDITIONS: Coagulopathy; Rethoracotomy; Blood Loss; Transfusion Requirements
Keywords: modified ultrafiltration; cardiac surgery; ROTEM; Multiple Electrode Aggregometry
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with modified ultrafiltration: elective cardiac surgery patients undergoing complex surgical intervention:
  coronary artery bypass grafting AND valve surgery double valve surgery aortic surgery Re-Dos
  Interventions: Device: modified ultrafiltration using Maquet haemoconcentrator, BC 20 plus
- without modified ultrafiltration: elective cardiac surgery patients undergoing complex surgical intervention:
  coronary artery bypass grafting AND valve surgery double valve surgery aortic surgery Re-Dos
  Interventions: Device: modified ultrafiltration using Maquet haemoconcentrator, BC 20 plus

INTERVENTIONS:
Device: modified ultrafiltration using Maquet haemoconcentrator, BC 20 plus — usage of modified ultrafiltration following extracorporeal circulation; filtration about 1,5 liters and re-fill with colloids
  Other Names: Maquet haemoconcentrator, BC 20 plus

SUMMARY:
The purpose of this study is to find out, whether filtration of the blood in patients undergoing cardiac surgery, beneficially influences the coagulation system.

DETAILED DESCRIPTION:
The impact of modified ultrafiltration following extracorporeal circulation on primary and secondary hemostasis is controversial. In this study we intend to assess both, primary and secondary hemostasis prior to and after the usage of modified ultrafiltration. Primary hemostasis is assessed using Multiple Electrode Aggregometry (Multiplate) and secondary hemostasis is assessed performing thrombelastometry using the ROTEM device. Patients are preoperatively randomized to receive either modified ultrafiltration or no filtration.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing complex cardiac surgery procedures

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: electice cardiac surgery patients undergoing complex procedures: CABG and valve double-valve aortic surgery Re-Dos
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
ex vivo platelet aggregation (TRAPtest) | 20 min after filtration

SECONDARY OUTCOMES:
secondary hemostasis assessed by ROTEM | 20 min before and after filtration
blood loss | 24 h after filtration
kind and number of transfused blood products | 24h after filtration
conventional coagulation analyses (INR, aPTT, platelet count, fibrinogen concentration) | 20 min before and after filtration
rate of rethoracotomy for bleeding | 24h after filtration

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Weber, Dr., Principal Investigator — Goethe University Frankfurt, Clinic for Anaesthesiology, Theodor Stern Kai 7, 60590 Frankfurt am Main, Germany
Locations (1):
- Goethe University hospital, Clinic for Anaesthesioloy, Frankfurt am Main, Germany

REFERENCES:
- [Background] Boodhwani M, Williams K, Babaev A, Gill G, Saleem N, Rubens FD. Ultrafiltration reduces blood transfusions following cardiac surgery: A meta-analysis. Eur J Cardiothorac Surg. 2006 Dec;30(6):892-7. doi: 10.1016/j.ejcts.2006.09.014. Epub 2006 Oct 13. PMID 17046273
- [Derived] Weber CF, Jambor C, Strasser C, Moritz A, Papadopoulos N, Zacharowski K, Meininger D. Normovolemic modified ultrafiltration is associated with better preserved platelet function and less postoperative blood loss in patients undergoing complex cardiac surgery: a randomized and controlled study. J Thorac Cardiovasc Surg. 2011 May;141(5):1298-304. doi: 10.1016/j.jtcvs.2010.09.057. Epub 2010 Dec 3. PMID 21130474